CLINICAL TRIAL: NCT00248261
Title: Effects of Ziprasidone vs. Placebo During the First Four Weeks of Eight Weeks Sertraline Treatment in Patients With Post-traumatic Stress Disorder (PTSD)
Brief Title: Ziprasidone and Sertraline in PTSD
Status: Terminated | Type: Observational
Why Stopped: High rate of early drop-outs
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: ZiSe; NRA1280017
Record Dates: First submitted 2005-11-02; First posted 2005-11-03 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Post-traumatic Stress Disorder
Keywords: ziprasidone, sertraline, PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — ziprasidone; Sertraline

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Drug: ziprasidone, sertraline

SUMMARY:
Serotonin re-uptake inhibitors, such as sertraline, are the medication of choice in post-traumatic stress disorder. However, it takes several weeks before they ameliorate symptoms. Therefore, we will add ziprasidone (vs. placebo) medication during the first four weeks of sertraline in order to find out if this strategy accelerates symptomatic relief.

DETAILED DESCRIPTION:
A current problem in the pharmacotherapy of PTSD is that the medication of choice, serotonin re-uptake inhibitors, take several weeks before they show considerable effects on PTSD symptoms. Addition of typical neuroleptics, such as ziprasidone, offers a potential strategy to bring about a faster symptomatic relief, because they display anxiolytic properties without the risk of dependence. Therefore, in addition to standard sertraline therapy (at least 8 weeks), we will give ziprasidone vs. placebo over the first four weeks in a double-blind randomized design.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Post-Traumatic Stress Disorder

Exclusion Criteria:

Lifetime psychotic disorders, current substance dependency, gravidity, lactation, tartrazine hypersensitivity, contraindication against sertraline or ziprasidone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PTSD patients
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2005-11; Primary Completion 2009-08 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Post-Traumatic Diagnostic Scale (PDS) | 56 days

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI) | 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Kellner, MD, PhD, Principal Investigator — UKE, Dep. of Pschiatry and Psychotherapy, Hamburg, Germany
Locations (1):
- UKE, Dept. of Psychiatry and Psychotherapy, Hamburg, Germany

REFERENCES:
- [Result] Kellner M, Muhtz C, Wiedemann K. Primary add-on of ziprasidone in sertraline treatment of posttraumatic stress disorder: lessons from a stopped trial? J Clin Psychopharmacol. 2010 Aug;30(4):471-3. doi: 10.1097/JCP.0b013e3181e79600. No abstract available. PMID 20631571